CLINICAL TRIAL: NCT05634681
Title: Plan-of-the-day Radiotherapy for Patients With Locally Advanced Cervical Cancer - a Prospective Randomized Controlled Trial (the POD-protocol)
Brief Title: Plan of the Day Radiotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Kjersti Bruheim, MD PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 236807
Record Dates: First submitted 2022-11-22; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Cervix Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental)
  Interventions: Radiation: Plan of the day
- Control arm (Active Comparator)
  Interventions: Radiation: Standard plan

INTERVENTIONS:
Radiation: Plan of the day — Several treatment plans are prepared and the appropriate plan is used at each treatment session.
  Arms: Intervention arm
Radiation: Standard plan — One treatment plan
  Arms: Control arm

SUMMARY:
The study objectives are to improve the treatment of LACC patients and to increase knowledge of the potential benefit of the plan-of-the-day concept on side effects during and after radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cervical cancer eligible for definitve radiochemotherapy
* FIGO stage IB1-IVa
* Over 18 years
* Speaks and understands Norwegian or English.
* ECOG 0-2
* Histology: Squamous cell carcinoma, adenocarcinoma, adenosquamous carcinoma
* Ability to understand and fill in patient questionnaires, and willing to sign a written informed consent
* Large movers (LM), fundus movement ≥2,5 cm.

Exclusion Criteria:

* Evidence of distant metastasis. Suspicious paraaortic lymphnodes below the renal vessels is allowed if they are covered by the radiation field
* Patients with previous surgery for their cervical cancer
* Uncontrolled intercurrent somatic illness.
* Psychiatric illness /social situations limiting study compliance
* Prior radiotherapy to the pelvis
* Patients who are pregnant or breastfeeding is excluded due to risk of teratogenic and abortifacient effects of radiotherapy and cisplatin, and the potential risk of adverse effect of nursing infants
* Patients under current treatment for other invasive s except non-melanoma skin cancers
* Nephrostomy
* Patients with inflammatory bowel disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2022-11-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
To investigate whether implementation of the plan of the day concept results in less gastro-intestinal toxicity. | 5 weeks
  To compare the change in patient reported acute diarrhea from baseline to week 4 from start of the treatment and to the end of external radiotherapy.
  Item 17 in EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Overall Officials: Kjersti Bruheim, MD PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway